CLINICAL TRIAL: NCT06379334
Title: Identification of Urinary Protein Biomarkers for Hepatocellular Carcinoma in Chronic Hepatitis B Patients
Brief Title: Discovering Urinary Protein Biomarkers for Hepatocellular Carcinoma in Chronic Hepatitis B Population
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-22PJ911
Record Dates: First submitted 2024-04-16; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCC: Urine samples from patients with chronic hepatitis B related hepatocellular carcinoma were collected and their proteomes were analyzed via liquid chromatography with tandem mass
  Interventions: Diagnostic Test: Urine test
- CHB: Urine samples from patients with chronic hepatitis B were collected and their proteomes were analyzed via liquid chromatography with tandem mass
  Interventions: Diagnostic Test: Urine test
- HC: Urine samples from healthy controls were collected and their proteomes were analyzed via liquid chromatography with tandem mass
  Interventions: Diagnostic Test: Urine test
- Other cancer: Urine samples from other cancer controls were collected and their proteomes were analyzed via liquid chromatography with tandem mass
  Interventions: Diagnostic Test: Urine test

INTERVENTIONS:
Diagnostic Test: Urine test — Urine samples were collected and their proteomes were analyzed via liquid chromatography with tandem mass spectrometry using data-dependent acquisition or parallel reaction monitoring.

SUMMARY:
Chronic hepatitis B (CHB) can lead to hepatocellular carcinoma (HCC), imposing a significant health and economic burden globally. Early detection of hepatitis B virus-related HCC (HBV-HCC) in CHB with potential biomarkers has become a pressing and difficult challenge. Recent advancements in urinary proteomics offer a promising approach for HBV-HCC biomarker identification, utilizing Liquid chromatography with tandem mass spectrometry for urine proteome analysis. Differential analysis using limma in R software will uncover upregulated proteins in HBV-HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old;
2. Previously healthy individuals without underlying diseases, confirmed to be free of hepatitis B infection through HBV serum markers, with regular physical examinations and blood biochemistry tests;
3. Chronic hepatitis B patients diagnosed through HBV serum markers, alpha-fetoprotein (AFP) concentration, clinical features, or imaging examinations;
4. Hepatitis B-related liver cancer patients with complete clinical data, preoperatively tested positive for HBsAg, diagnosed based on clinical features and imaging examinations preoperatively, and pathologically confirmed with HCC postoperatively;
5. Patients with non-hepatocellular liver cancer, preoperatively diagnosed based on clinical features and imaging examinations, with negative HBsAg, and pathologically or by biopsy confirmed as non-hepatocellular liver cancer without liver metastasis, with complete clinical data and no liver metastasis;
6. Able to independently sign an informed consent form.

Exclusion Criteria:

1. Patients with long-term heavy alcohol consumption;
2. Patients with chronic hepatitis C infection;
3. Patients with autoimmune diseases;
4. Patients who have taken drugs known to have definite hepatotoxicity within the past year;
5. Patients with urinary system infections;
6. Patients with hematuria;
7. Patients with significant proteinuria;
8. Patients with tumors of the urinary system;
9. Patients with acute infectious diseases;
10. Patients with hepatitis B-related liver cancer who also have tumors other than primary hepatocellular carcinoma.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age > 18 years old;
  2. Previously healthy individuals without underlying diseases, confirmed to be free of hepatitis B infection through HBV serum markers, with regular physical examinations and blood biochemistry tests;
  3. Chronic hepatitis B patients diagnosed through HBV serum markers, AFP concentration, clinical features, or imaging examinations;
  4. Hepatitis B-related liver cancer patients with complete clinical data, preoperatively tested positive for HBsAg, diagnosed based on clinical features and imaging examinations preoperatively, and pathologically confirmed with HCC postoperatively;
  5. Patients with non-hepatocellular liver cancer, preoperatively diagnosed based on clinical features and imaging examinations, with negative HBsAg, and pathologically or by biopsy confirmed as non-hepatocellular liver cancer without liver metastasis, with complete clinical data and no liver metastasis;
  6. Able to independently sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-12-06 (Actual); Primary Completion 2024-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
upregulated proteins | 2024-5
downregulated proteins | 2024-5

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No